CLINICAL TRIAL: NCT05622058
Title: A Phase 1b Clinical Study of the Dual MDMX/MDM2 Inhibitor, ALRN-6924, as a Chemoprotection Agent in Patients With TP53-Mutated, HER2 Negative Breast Cancer Receiving Neoadjuvant or Adjuvant Chemotherapy With Docetaxel, Doxorubicin, and Cyclophosphamide (TAC)
Brief Title: A Study of ALRN-6924 for Protection of Chemotherapy-Induced Side Effects in Patients With TP53-Mutant Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study has been terminated early given that the first four patients enrolled have experienced Grade 4 neutropenia and alopecia after cycle 1 and as such failed to meet the primary endpoint and the main secondary endpoint.
Sponsor: Aileron Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ALRN-6924-1-05; 2022-000158-27 (EudraCT Number)
Record Dates: First submitted 2022-06-01; First posted 2022-11-18 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Prevention of Chemotherapy-induced Myelosuppression
Keywords: ALRN-6924; Chemoprotection; Myelosuppression; Cell cycle arrest; p53 mutation; Breast cancer; Alopecia; Neutropenia
MeSH Terms: conditions — Breast Neoplasms; Alopecia; Neutropenia | interventions — Doxorubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALRN-6924 Dose plus TAC (Experimental): ALRN-6924 plus Docetaxel, Doxorubicin, and Cyclophosphamide (TAC)
  Interventions: Drug: ALRN-6924; Drug: TAC (doxorubicin 50 mg/m2; cyclophosphamide 500 mg/m2; docetaxel 75 mg/m2)

INTERVENTIONS:
Drug: ALRN-6924 — ALRN-6924 administered in every chemotherapy treatment cycle as an IV infusion over 1 hour on Days 0 (approximately 18 hours prior to chemotherapy administration), 1 (approximately 1 hour prior to chemotherapy administration), and 2 (approximately 24 hours after the second infusion of ALRN-6924).
Drug: TAC (doxorubicin 50 mg/m2; cyclophosphamide 500 mg/m2; docetaxel 75 mg/m2) — TAC will be administered as an IV infusion on Day 1 of every 3-week treatment cycle

SUMMARY:
This is a Phase 1b open-label, single arm, multicenter, study of ALRN-6924 as a chemoprotection agent in patients with TP53-mutated HER2- breast cancer (stages IIa to IIIb) receiving neoadjuvant or adjuvant chemotherapy with doxorubicin, docetaxel, and cyclophosphamide (TAC). Chemotherapy affects cells that are dividing, whether they are tumor cells or healthy cells (including, bone marrow cells, hair follicle cells, and epithelial cells lining the gastrointestinal tract). ALRN-6924 is designed to stop cell division in healthy cells but not in tumor cells because they have a mutation of the TP53 gene. When this happens, tumor cells will still be destroyed by the chemotherapy but healthy cells that are not dividing may be spared from chemotherapy damage and the patient should have less side effects.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, single-arm, multicenter clinical trial for evaluation of safety, tolerability and chemoprotection effects of ALRN-6924 combined with chemotherapy in patients with TP53-mutated, HER2 negative breast cancer without distant organ metastases. All patients will receive the neoadjuvant or adjuvant chemotherapy regimen known as TAC. TAC consists of doxorubicin 50 mg/m2 IV infusion, docetaxel 75mg/m2 IV infusion and cyclophosphamide 500 mg/m2 IV infusion, given on Day 1 of every 3-week cycle for a total of 4-6 treatment cycles according to each patient's individual needs, individual institutional policies and standards of care, as well as investigator discretion. ALRN-6924 1.2 mg/kg will be administered on 3 consecutive days in each treatment cycle, Days 0-2. Prophylactic administration of G-CSF prior to the first instance of Grade 4 neutropenia is not allowed in Cycle 1. Myeloid growth factor support with filgrastim should be administered immediately if a patient is diagnosed with Grade 4 neutropenia.

ELIGIBILITY:
Inclusion Criteria:

* Females and males, age ≥18years.
* Patients who, in the investigator's judgment, are able to understand and willing to comply with the requirements of this clinical trial and to provide written informed consent.
* Histologically confirmed diagnosis of HER2 negative breast cancer
* Candidate to receive chemotherapy with TAC regimen
* Presence of p53 mutation(s) in tumor tissue as assessed by next generation sequencing (NGS).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤2
* Left ventricular ejection fraction > 55%.
* Laboratory results obtained within 14 days prior to the first study treatment administration (Cycle 1, Day 0) demonstrating:

  * Absolute neutrophil count (ANC) ≥ 1500 cells/μL (without granulocyte colony stimulating factor [G-CSF] support within 2 weeks prior to the first study treatment administration)
  * Platelet count ≥ 100,000/μL (without transfusion within 2 weeks prior to the first study treatment administration)
  * Hemoglobin ≥ 10.0 g/dL
  * AST, ALT, and alkaline phosphatase ≤ 2.5 x the upper limit of normal (ULN)
  * Serum bilirubin ≤ 1.5× ULN (patients with known Gilbert's disease who have serum bilirubin level ≤ 3× ULN may be enrolled.)
  * Patients who are not receiving therapeutic anticoagulation: Calculated creatinine clearance (CrCl) ≥ 30 mL/min (Cockcroft-Gault formula).
* Have not received prior chemotherapy or targeted systemic therapy for their breast cancer.

Exclusion Criteria:

* Known hypersensitivity to any component of study treatment.
* Prior chemotherapy for HER2 negative breast cancer.

  1. Presence of distant metastases. Nodal involvement is acceptable.
* Uncontrolled intercurrent illness including but not limited to:

  * Clinically significant, active, uncontrolled infection including human immunodeficiency virus (HIV), or hepatitis B or C

    * Patients with HIV must be on effective antiretroviral therapy for ≥ 4 weeks prior to enrollment and have HIV viral load < 400 copies/mL, have had no acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections in the past 12 months, and have CD4+ count ≥ 350 cells/μL.
    * Patients with chronic hepatitis B virus (HBV) must be on antiviral therapy and have HBV viral load below the limits of detection.
    * Patients with hepatitis C virus (HCV) must be on or have completed antiviral therapy and have an HCV viral load below the limits of detection.
  * Uncontrolled hypertension
  * Uncontrolled diabetes mellitus
* Clinically unstable cardiac disease, including unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, active myocardial ischemia, or indwelling temporary pacemaker.
* Pregnant or lactating women.
* Hereditary angioedema of any severity or severe or life-threatening angioedema due to any cause.
* Treatment with an investigational agent for any indication within the shorter of 14 days or 5 half-lives, if the half-life is known.
* The required use of any concomitant medications that are predominantly cleared by hepatobiliary transporters, OATP members OATP1B1 and OATP1B3, on the day of the first ALRN-6924 infusion to within 48 hours after the last ALRN-6924 infusion in a treatment cycle. This criterion does not apply to the patients in the control group.
* Other medications, severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
* Clinically evident alopecia of any grade at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ALRN-6924 in combination with TAC chemotherapy | Approximately 24 weeks
  Proportion of patients with Common Terminology Criteria for Adverse Events (CTCAE) Grade 3/4 treatment emergent adverse events (TEAEs); proportion of patients with treatment-related adverse events and serious adverse events as assessed by NCI CTCAE v5.0
  Clinical and laboratory adverse events (AEs) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). System Organ Class (SOC) and Preferred Term (PT) will be attached to the clinical database. AE severity will be graded using the CTCAE.
  All AEs will be summarized (incidence) and listed by the System Organ Class (SOC), preferred term, toxicity/severity grade, and causal relationship to study medication. In addition, separate summaries of SAEs and Grade 3 and 4 AEs will be presented.
Chemoprotective effects of ALRN-6924 on bone marrow toxicities | Approximately 3 weeks for each patient
  Incidence and duration of Grade 4 neutropenia in Cycle 1
  for each treatment cycle and all cycles combined

SECONDARY OUTCOMES:
Chemoprotective effects of ALRN-6924 on alopecia induced by TAC | Approximately 24 weeks
  Incidence of Grade 2 alopecia after treatment with ALRN-6924 plus TAC
Chemoprotective effects of ALRN-6924 on neutropenia | Approximately 24 weeks
  Incidence rate of grade 4 neutropenia for each treatment cycle and all cycles combined
Time to absolute neutrophil count (ANC) recovery in Cycle 1 | 3 weeks (cycle 1)
  Time in days from ANC nadir to recovery
Depth of ANC nadir in Cycle 1 | 3 weeks (cycle 1)
  Lowest ANC count during cycle 1
Chemoprotective effects of ALRN-6924 on Grade ≥3 neutropenia for each cycle and all cycles | Approximately 24 weeks
  CTCAE v5 grade 3 neutropenia
Chemoprotective effects of ALRN-6924 on thrombocytopenia | Approximately 24 weeks
  CTCAE v5 grade ≥3 thrombocytopenia
Chemoprotective effects of ALRN-6924 on anemia | Approximately 24 weeks
  CTCAE v5 grade ≥3 anemia
Chemoprotective effects of ALRN-6924 on febrile neutropenia | Approximately 24 weeks
  Incidence of febrile neutropenia for each cycle and all cycles
Chemoprotective effects of ALRN-6924 on the need for chemotherapy dose reductions | Approximately 24 weeks
  Number of dose reductions of chemotherapy due to chemotherapy-related toxicity for each cycle and all cycles
Use of myeloid growth factors | Approximately 24 weeks
  Number of instances of granulocyte colony-stimulating factors (G-CSF) use to treat Grade 4 neutropenia for each cycle and all cycles
Need for red blood cell transfusions | Approximately 24 weeks
  Number of red blood cell (RBC) transfusions during each cycle and all cycles
Need for platelet transfusions | Approximately 24 weeks
  Number of platelet transfusions during each cycle and all cycles
  The ALRN-6924 PK profile with and without AC chemotherapy will be compared.
PK of ALRN-6924 | Cycle 1 (each cycle is 21 days)
  PK parameters (e.g., area-under-the-curve [AUC]) of ALRN-6924
PK of ALRN-6924 | Cycle 1 (each cycle is 21 days)
  PK parameters (e.g., maximum concentration [Cmax] of ALRN-6924
PK of ALRN-6924 | Cycle 1 (each cycle is 21 days)
  PK parameters (e.g., time of Cmax [tmax]) of ALRN-6924
PK of ALRN-6924 | Cycle 1 (each cycle is 21 days)
  PK parameters (e.g., half-life [t1/2]) of ALRN-6924
Efficacy of chemotherapy | Approximately 24 weeks
  Tumor response after TAC chemotherapy: proportion of patients with pCR after completion of neoadjuvant chemotherapy and surgery, per local standard of care and institutional policies

CONTACTS AND LOCATIONS:
Locations (14):
- United States (5):
  - Oncology and Hematology Associates of West Broward, Tamarac, Florida
  - Southern Oncology Specialists, Huntersville, North Carolina
  - Regional Medical Oncolgy Center, Wilson, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Pennsylvania Cancer Specialists & Resesrach Institute, Gettysburg, Pennsylvania
- Bosnia and Herzegovina (4):
  - University Clinical Center of the Republic of Srpska, Banja Luka
  - University Clinical Hospital Mostar, Mostar
  - Clinical Center University of Sarajevo, Oncology Clinic, Sarajevo
  - University Clinical Center Tuzla, Tuzla
- Bulgaria (2):
  - MBAL University Hospital OOD, Panagyurishte
  - KOC (Complex Oncology Center) Plovdiv, Plovdiv
- Serbia (3):
  - Kliničko bolnički centar "Bežanijska kosa", Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
  - Univerzitetski Klinički centar Kragujevac, Kragujevac